CLINICAL TRIAL: NCT02650531
Title: Norwegian COgnitive Impairment After STroke (NorCOAST) Study
Acronym: Nor-Coast
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Ullevaal University Hospital (Other); Vestre Viken Hospital Trust (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/171/REK nord
Record Dates: First submitted 2015-12-10; First posted 2016-01-08 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Dementia; Mild Cognitive Impairment; Stroke
Keywords: Follow up studies; Risk factors
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective observational multicenter study aiming to describe incidence, and identify predictors for development of poststroke dementia (PSD) and mild cognitive impairment (MCI) after stroke

DETAILED DESCRIPTION:
About 15000 Norwegians suffer a stroke every year and 2/3 will be more or less disabled. In addition to motor impairments and comorbidities, disability after stroke is often related to post stroke dementia (PSD) or mild neurocognitive disorder (NCD). However, these problems are hardly addressed in stroke or dementia research and frequently ignored in clinical practise. In the Nor-COAST study an interdisciplinary research group will collaborate to establish a research platform across all Norwegian Health Authorities. The overall aim of the study is to improve competence on PSD and NCD in order to improve individual health outcomes following a stroke. The specific objectives are to determine the incidence of PSD and NCD and the consequences on function and use of health care services and to enhance the early detection of PSD and NCD by identifying a set of risk factors, ranging from genetics to physical activity. The incidence and impact of PSD and NCD on function and use of health care services, medication and life-style changes are important when planning future health care services. Tools identifying patients at risk might improve diagnostic work up and together with knowledge on pathogenic aspects it will contribute to future treatment and prevention of PSD and NCD.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis according to the WHO criteria

Exclusion Criteria:

* Not scandinavian speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute stroke
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
Score on the Montreal cognitive assessment (MOCA) | 18 months
  Performance based test

SECONDARY OUTCOMES:
Score on the Montreal cognitive assessment (MOCA) | 3 months
  Performance based test
Time spent in upright position | 3 months
  measured by bodyworn sensors
Time spent in upright position | 18 months
  measured by bodyworn sensors
Brain Imaging | 18 months
  MRI
Score on Short Physical Performance Battery (sppb) | 3 months
  Performance based test for mobility and lower extremity function
Score on Short Physical Performance Battery (sppb) | 18 months
  Physical function by performance based tests
Selfreported habits concerning smoking, alcohol, diet and medication using standardised questionnaires | 3 months
Selfreported habits concerning smoking, alcohol, diet and medication using standardised questionnaires | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, md prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Thingstad P, Askim T, Beyer MK, Brathen G, Ellekjaer H, Ihle-Hansen H, Knapskog AB, Lydersen S, Munthe-Kaas R, Naess H, Pendlebury ST, Seljeseth YM, Saltvedt I. The Norwegian Cognitive impairment after stroke study (Nor-COAST): study protocol of a multicentre, prospective cohort study. BMC Neurol. 2018 Nov 26;18(1):193. doi: 10.1186/s12883-018-1198-x. PMID 30477436
- [Result] Waehler IS, Saltvedt I, Lydersen S, Fure B, Askim T, Einstad MS, Thingstad P. Association between in-hospital frailty and health-related quality of life after stroke: the Nor-COAST study. BMC Neurol. 2021 Mar 4;21(1):100. doi: 10.1186/s12883-021-02128-5. PMID 33663430
- [Derived] Sandvig HV, Saltvedt I, Edwin TH, Aam S, Alme KN, Eldholm RS, Lydersen S, Mollnes TE, Munthe-Kaas R, Ueland PM, Ulvik A, Wethal T, Knapskog AB. Associations between systemic inflammation and cognitive trajectories post-stroke. Sci Rep. 2025 Nov 28;15(1):42791. doi: 10.1038/s41598-025-27119-1. PMID 41315409
- [Derived] Sandvig HV, Aam S, Alme KN, Lydersen S, Magne Ueland P, Ulvik A, Wethal T, Saltvedt I, Knapskog AB. Neopterin, kynurenine metabolites, and indexes related to vitamin B6 are associated with post-stroke cognitive impairment: The Nor-COAST study. Brain Behav Immun. 2024 May;118:167-177. doi: 10.1016/j.bbi.2024.02.030. Epub 2024 Feb 28. PMID 38428649
- [Derived] Luzum G, Thrane G, Aam S, Eldholm RS, Grambaite R, Munthe-Kaas R, Thingstad P, Saltvedt I, Askim T. A Machine Learning Approach to Predict Post-stroke Fatigue. The Nor-COAST study. Arch Phys Med Rehabil. 2024 May;105(5):921-929. doi: 10.1016/j.apmr.2023.12.005. Epub 2024 Jan 17. PMID 38242298
- [Derived] Navickaite E, Saltvedt I, Lydersen S, Munthe-Kaas R, Ihle-Hansen H, Grambaite R, Aam S. Diagnostic accuracy of the Clock Drawing Test in screening for early post-stroke neurocognitive disorder: the Nor-COAST study. BMC Neurol. 2024 Jan 9;24(1):22. doi: 10.1186/s12883-023-03523-w. PMID 38195396
- [Derived] Luzum G, Gunnes M, Lydersen S, Saltvedt I, Tan X, Thingstad P, Thrane G, Askim T. Physical Activity Behavior and Its Association With Global Cognitive Function Three Months After Stroke: The Nor-COAST Studydagger. Phys Ther. 2023 Dec 6;103(12):pzad092. doi: 10.1093/ptj/pzad092. PMID 37440440
- [Derived] Sandvig HV, Aam S, Alme KN, Askim T, Beyer MK, Ellekjaer H, Ihle-Hansen H, Lydersen S, Mollnes TE, Munthe-Kaas R, Naess H, Saltvedt I, Seljeseth YM, Thingstad P, Wethal T, Knapskog AB. Plasma Inflammatory Biomarkers Are Associated With Poststroke Cognitive Impairment: The Nor-COAST Study. Stroke. 2023 May;54(5):1303-1311. doi: 10.1161/STROKEAHA.122.041965. Epub 2023 Apr 7. PMID 37026459
- [Derived] Gynnild MN, Hageman SHJ, Spigset O, Lydersen S, Saltvedt I, Dorresteijn JAN, Visseren FLJ, Ellekjaer H. Use of lipid-lowering therapy after ischaemic stroke and expected benefit from intensification of treatment. Open Heart. 2022 Apr;9(1):e001972. doi: 10.1136/openhrt-2022-001972. PMID 35459718
- [Derived] Munthe-Kaas R, Aam S, Saltvedt I, Wyller TB, Pendlebury ST, Lydersen S, Hagberg G, Schellhorn T, Rostoft S, Ihle-Hansen H. Is Frailty Index a better predictor than pre-stroke modified Rankin Scale for neurocognitive outcomes 3-months post-stroke? BMC Geriatr. 2022 Feb 19;22(1):139. doi: 10.1186/s12877-022-02840-y. PMID 35183106
- [Derived] Einstad MS, Thingstad P, Lydersen S, Gunnes M, Saltvedt I, Askim T. Physical Performance and Cognition as Predictors of Instrumental Activities of Daily Living After Stroke: A Prospective Multicenter Cohort Study. Arch Phys Med Rehabil. 2022 Jul;103(7):1320-1326. doi: 10.1016/j.apmr.2022.01.153. Epub 2022 Feb 16. PMID 35181266
- [Derived] Alme KN, Ulvik A, Askim T, Assmus J, Mollnes TE, Naik M, Naess H, Saltvedt I, Ueland PM, Knapskog AB. Neopterin and kynurenic acid as predictors of stroke recurrence and mortality: a multicentre prospective cohort study on biomarkers of inflammation measured three months after ischemic stroke. BMC Neurol. 2021 Dec 8;21(1):476. doi: 10.1186/s12883-021-02498-w. PMID 34879833
- [Derived] Alme KN, Askim T, Assmus J, Mollnes TE, Naik M, Naess H, Saltvedt I, Ueland PM, Ulvik A, Knapskog AB. Investigating novel biomarkers of immune activation and modulation in the context of sedentary behaviour: a multicentre prospective ischemic stroke cohort study. BMC Neurol. 2021 Aug 16;21(1):318. doi: 10.1186/s12883-021-02343-0. PMID 34399717
- [Derived] Schellhorn T, Zucknick M, Askim T, Munthe-Kaas R, Ihle-Hansen H, Seljeseth YM, Knapskog AB, Naess H, Ellekjaer H, Thingstad P, Wyller TB, Saltvedt I, Beyer MK. Pre-stroke cognitive impairment is associated with vascular imaging pathology: a prospective observational study. BMC Geriatr. 2021 Jun 14;21(1):362. doi: 10.1186/s12877-021-02327-2. PMID 34126944
- [Derived] Schellhorn T, Aamodt EB, Lydersen S, Aam S, Wyller TB, Saltvedt I, Beyer MK. Clinically accessible neuroimaging predictors of post-stroke neurocognitive disorder: a prospective observational study. BMC Neurol. 2021 Feb 25;21(1):89. doi: 10.1186/s12883-021-02117-8. PMID 33632149
- [Derived] Einstad MS, Saltvedt I, Lydersen S, Ursin MH, Munthe-Kaas R, Ihle-Hansen H, Knapskog AB, Askim T, Beyer MK, Naess H, Seljeseth YM, Ellekjaer H, Thingstad P. Associations between post-stroke motor and cognitive function: a cross-sectional study. BMC Geriatr. 2021 Feb 5;21(1):103. doi: 10.1186/s12877-021-02055-7. PMID 33546620
- [Derived] Munthe-Kaas R, Aam S, Saltvedt I, Wyller TB, Pendlebury ST, Lydersen S, Ihle-Hansen H. Test Accuracy of the Montreal Cognitive Assessment in Screening for Early Poststroke Neurocognitive Disorder: The Nor-COAST Study. Stroke. 2021 Jan;52(1):317-320. doi: 10.1161/STROKEAHA.120.031030. Epub 2020 Nov 30. PMID 33250039
- [Derived] Alme KN, Knapskog AB, Naess H, Naik M, Beyer M, Ellekjaer H, English C, Hansen HI, Kummeneje CS, Munthe-Kaas R, Saltvedt I, Seljeseth Y, Tan X, Thingstad P, Askim T. Is long-bout sedentary behaviour associated with long-term glucose levels 3 months after acute ischaemic stroke? A prospective observational cohort study. BMJ Open. 2020 Nov 26;10(11):e037475. doi: 10.1136/bmjopen-2020-037475. PMID 33243789
- [Derived] Gynnild MN, Aakeroy R, Spigset O, Askim T, Beyer MK, Ihle-Hansen H, Munthe-Kaas R, Knapskog AB, Lydersen S, Naess H, Rosstad TG, Seljeseth YM, Thingstad P, Saltvedt I, Ellekjaer H. Vascular risk factor control and adherence to secondary preventive medication after ischaemic stroke. J Intern Med. 2021 Mar;289(3):355-368. doi: 10.1111/joim.13161. Epub 2020 Aug 19. PMID 32743852